CLINICAL TRIAL: NCT06169007
Title: Role of Soluble Immune Checkpoints Molecules as Diagnostic and Prognostic Markers in Breast Cancer Patients
Brief Title: Using of Costimulatory and co Inhibatory Immune Checkpoints as Diagnostic and Prognostic in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Soliman Khalfallah, Principal investigator, Assiut University
Other Study IDs: Immune checkpoints in cancer
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: breast cancer and sCD40 and sTIM-3
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Checkpoint proteins regulate the immune system; breast cancer cells exploit the up-regulation or down-regulation of these proteins to evade anti-tumour immune responses . It is now well recognized that advanced metastatic BC and early disease are associated with both localized and systemic immune dysfunction .in this study levels of soluble immune checkpoint molecules sTIM3 and sCD40 will be measured and compared with tissue form ,then follow up to patients' prognosis and the relation to markers levels.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumour and the leading cause of cancer-associated mortality among women .Although comprehensive therapies exist, patient response to the treatments significantly varies, which partly attributed to varying antitumor immune responses .Immunotherapy is being recognized as a key therapeutic modality for cancer and represents one of the most promising therapies. Checkpoint proteins regulate the immune system. Breast cancer (BC) cells exploit the up-regulation or down-regulation of these proteins to evade anti-tumour immune responses. Notwithstanding the existence of profound immune dysregulation in advanced metastatic breast cancer (BC), it is now well recognized that early disease is also associated with both localized and systemic immune dysfunction . Recently, soluble co-inhibitory immune checkpoint molecules (ICMs) have been implicated as being potential mediators of the systemic immune dysregulation . Prominent among these soluble co inhibitory ICMs are: cytotoxic T-lymphocyte-associated protein (CTLA-4), programmed cell death protein 1 (PD-1) and its ligand, PD-L1, lymphocyte activation gene 3 (LAG-3) and T- Cell immunoglobulin and mucin-domain-containing protein 3 (TIM-3) . A study showed that resistance to anti-CTLA-4 or anti PD-1/PD-L1 inhibitors is compensated by up regulation of other immune checkpoints, such as Tim-3 . Consequently, Tim-3 has gained prominence as a potential candidate for cancer immunotherapy. Blocking Tim-3 with other checkpoint inhibitors has been shown to enhance antitumor immunity and suppress tumour growth in several preclinical tumour models. Increasing numbers of novel receptors and ligands have recently been found in the immune system. Some take part in a costimulatory interactions, such as Glucocorticoid-induced TNFR-related protein (GITR), GITR Ligand, CD27, CD28, CD40, CD80, CD86 and Inducible Co-Stimulator (ICOS) . CD40-CD40 ligand (CD40L) pathway is a member of the TNF superfamily and is expressed at various levels on antigen-presenting cells, epithelial cells, and hematopoietic progenitor cells . The CD40-CD40L costimulatory pathway has been shown to play a crucial role in humoral responses in humans, these cytokines modulate the function of T lymphocytes in antitumor responses. Few Review studies have reported the levels of sTIM-3 and CD40 in the literature, we are going to assess them and compare different stages of breast cancer .Previous study reported that, the level of Plasma concentration of the co-stimulatory immune checkpoint CD40 as well as the co-inhibitory molecule TIM-3 were all significantly lower in early breast cancer patients compared to healthy controls. Following neoadjuvant chemotherapy NAC, the plasma concentrations of the soluble co-stimulatory ICM sCD40 and soluble co inhibitory ICM sTIM-3 were significantly increased

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer aged > 18 years attending the Medical Oncology department of South Egypt Cancer Institute

Exclusion Criteria:

* Patients on chemotherapy
* A history of any other malignancy
* known (HIV) and/or hepatitis B or hepatitis C viruses,
* pregnancy or breast feeding
* patients or controls that refuse to be a part of the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with breast cancer and healthy females as controls
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the levels of sTIM-3 and sCD40 in breast cancer patients in different stages and follow up their role in disease prognosis compared with healthy controls. Results will be compared with the previous studies. | study will take about 12months to be completed

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Fadel, lecturer, Study Director — Assiut University